CLINICAL TRIAL: NCT06598631
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Investigate the Efficacy and Safety of Volenrelaxin in Adults With Chronic Kidney Disease
Brief Title: Efficacy and Safety of Volenrelaxin in Adults With Chronic Kidney Disease
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to a lack of foreseeable clinical benefit in the proposed chronic kidney disease population, following the termination of a related heart failure study that demonstrated no benefit in an overlapping patient group.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18839; J3E-MC-EZDC (Other: Eli Lilly and Company); 2024-513895-16-00 (EU CTIS Number)
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Chronic Kidney Disease
Keywords: eGFR; UACR
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Volenrelaxin Dose 1 (Experimental): Participants will receive Volenrelaxin subcutaneously (SC)
  Interventions: Drug: Volenrelaxin
- Volenrelaxin Dose 2 (Experimental): Participants will receive Volenrelaxin SC
  Interventions: Drug: Volenrelaxin
- Volenrelaxin Dose 3 (Experimental): Participants will receive Volenrelaxin SC
  Interventions: Drug: Volenrelaxin
- Placebo (Placebo Comparator): Participants will receive Placebo SC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Volenrelaxin — Administered SC
  Other Names: LY3540378
  Arms: Volenrelaxin Dose 1; Volenrelaxin Dose 2; Volenrelaxin Dose 3
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study is to investigate the efficacy and safety of Volenrelaxin in adults with Chronic Kidney Disease. The study will last about 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of Chronic Kidney Disease (CKD) based on eGFR category and albuminuria category per the Kidney Disease: Improving Global Outcomes (KDIGO) criteria
* Have been on a maximally tolerated labeled daily dose of an angiotensin-converting enzyme inhibitor (ACEi) or an angiotensin receptor blocker (ARB) for 90 days preceding screening and is expected to remain on a stable regimen through the study
* If on additional treatment for CKD, must be on stable dose for at least 90 days before screening.
* If diagnosed with Type 2 Diabetes, should be on stable antihyperglycemic treatment for at least 90 days before screening.

Exclusion Criteria:

* Have any one of the following cardiovascular conditions 90 days prior to screening:

  * myocardial infarction
  * stroke
  * hospitalization or urgent visit for heart failure, and
  * coronary, carotid, or peripheral artery revascularization.
* Have a documented New York Heart Association (NYHA) Class IV heart failure at the time of screening.
* Have chronic or intermittent hemodialysis or peritoneal dialysis 90 days prior to screening.
* Have acute dialysis or acute kidney injury 90 days prior to screening.
* Have a history of a congenital or hereditary kidney disease, polycystic kidney disease, lupus nephritis, anti-neutrophil cytoplasmic antibody (ANCA)-associated vasculitis, and nephrotic syndrome
* Requires chronic immunosuppression.
* Have HbA1c >8.5% at screening
* Have had a transplanted organ or are awaiting an organ transplant
* Have a diagnosis or history of malignant disease within 5 years prior to baseline.
* Have symptomatic hypotension.
* Have acute or chronic hepatitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-10-09 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Percent Change from Baseline of Urine Albumin-Creatinine Ratio (UACR) | Baseline, Week 12

SECONDARY OUTCOMES:
Change from Baseline in Estimated Glomerular Filtration Rate (eGFR) | Baseline, Week 12
  Calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) creatinine equation [2009]
Change from Baseline in eGFR | Baseline, Week 12
  Calculated using the CKD-EPI creatinine equation [2021]

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (35):
- United States (16):
  - Rancho Research Institute, Downey, California
  - Southwest Nephrology Associates, Evergreen Park, Illinois
  - Nephrology Associates of Northern Illinois and Indiana (NANI) - Hinsdale, Hinsdale, Illinois
  - Nephrology Associates of Northern Illinois and Indiana (NANI) - Huntley, Huntley, Illinois
  - Nephrology Associates of Northern Illinois and Indiana (NANI) - Fort Wayne, Fort Wayne, Indiana
  - Nephrology Associates of Northern Illinois and Indiana - IKS - Indianapolis South, Indianapolis, Indiana
  - Diabetes and Metabolism Associates, APMC, Metairie, Louisiana
  - Elite Clinical Research Center, Flint, Michigan
  - Eastern Nephrology Associates - Greenville, Greenville, North Carolina
  - Eastern Nephrology Associates, Jacksonville, North Carolina
  - Eastern Nephrology Associates- Kinston Office, Kinston, North Carolina
  - Lucas Research, Inc., Morehead City, North Carolina
  - Eastern Nephrology Associates- New Bern Office, New Bern, North Carolina
  - Eastern Nephrology Associates - Wilmington, Wilmington, North Carolina
  - Endocrine Associates, Houston, Texas
  - Permian Research Foundation, Odessa, Texas
- Australia (4):
  - Renal Research - Gosford, Gosford, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - The Royal Melbourne Hospital, Parkville, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- China (6):
  - Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Taian City Central Hospital, Taian, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Ningbo 2nd Hospital, Ningbo, Zhejiang
  - The first affiliated hospital of Ningbo university, Ningbo, Zhejiang
- Japan (3):
  - Takai Internal Medicine Clinic, Kamakura-shi, Kanagawa
  - Niigata University Medical & Dental Hospital, Niigata
  - Okayama University Hospital, Okayama
- Spain (6):
  - CHUAC-Complejo Hospitalario Universitario A Coruña, A Coruña, A Coruña [La Coruña]
  - Hospital Universitario Virgen de la Victoria, Málaga, Andalusia
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [Barcelona]
  - Hospital Ribera Polusa, Lugo, Lugo [Lugo]
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid, Comunidad de
  - Hospital Clinico de Valencia, Valencia, Valenciana, Comunitat

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: Efficacy and Safety of Volenrelaxin in Adults with Chronic Kidney Disease — https://trials.lilly.com/en-US/trial/533476